CLINICAL TRIAL: NCT04264845
Title: Patient-Reported Outcomes as an Indicator of Disease Transitions in Heart Failure
Acronym: PRO-HF
Status: Active, not recruiting | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1050750
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Provider Focus Group: All heart failure providers at the participating centers will be screened as potential participants.
  Interventions: Other: Provider Focus
- Patient Interview Group: Patients with heart failure who are seen in the heart failure outpatient clinics at the participating centers will be screened for this study. The Principal Investigator will confirm the presence of heart failure based on established and agreed criteria. A real world, diverse population ranging from patients with milder forms of HF to the most advanced disease will be included in this study and allow the researchers to validate the prognostic models in larger, regionally diverse populations to better define the comparative effectiveness of alternative treatments in patients with different risk profiles.
  Interventions: Other: Patient Interview
- PROs/Clinical Data Integration Group: Patients with heart failure who are seen in the heart failure outpatient clinics at the participating centers will be screened for this study. The Principal Investigator will confirm the presence of heart failure based on established and agreed criteria. A real world, diverse population ranging from patients with milder forms of HF to the most advanced disease will be included in this study and allow the researchers to validate the prognostic models in larger, regionally diverse populations to better define the comparative effectiveness of alternative treatments in patients with different risk profiles.
  This group includes a sub-study of patients providing blood samples.
  Interventions: Other: PROs/Clinical Data Integration

INTERVENTIONS:
Other: Provider Focus — The provider focus groups will be conducted and data from the focus group sessions will be analyzed and used to evaluate clinicians' interpretation of PROs and acceptability of PRO data in routine clinical care. A formal provider training program will be designed and implemented by a subject matter expert. The focus group session will be repeated at 12 months, with the 12month administration having an increased emphasis on barriers, facilitators, and value of PROs in clinical care.
  Groups: Provider Focus Group
Other: Patient Interview — A trained professional interviewer will conduct a one-time, one-hour, semi-structured telephone interview of each subject to better understand patient experiences with HF, the treatment process and quality of life determinants. Two semistructured interviews will be conducted with the first 30 patients who have had LVAD therapy (of the 100 patients who agreed to be interviewed), before and 12 months after device implantation. The goal of these interviews will be to describe patient experiences with LVAD therapy, examine factors influencing quality of life, and determine whether currently available PRO tools are likely to capture the intended experiences in HF as they relate to LVAD therapy.
  Groups: Patient Interview Group
Other: PROs/Clinical Data Integration — A plan has been developed that will integrate PRO scores into patient medical records. Information will be obtained from 2 instruments (KCCQ12 and NIH PROMIS) that are routinely administered as part standard of care. PRO and clinical data will be obtained from electronic medical records of patients seen in the heart failure clinic. All required information will be obtained from the subjects' electronic medical records over a period of 3.5 years after enrollment into the study.
  Groups: PROs/Clinical Data Integration Group

SUMMARY:
This is a prospective, observational, open study that will utilize the following tools: survey/questionnaire research, interviews, and focus groups, and secondary/archival data analysis. In addition, a subset of selected subjects will be asked to provide blood samples to examine the biologic determinants of patient health status in heart failure (HF). This will help us understand better the biomarkers or genetic factors that may cause differences in patient quality of life.

DETAILED DESCRIPTION:
The primary endpoint of this study is the determination of the feasibility and efficiency of integrating routine PRO assessments into the clinical care of patients treated for HF. To reach this, three groups will be involved in the study.

Provider Focus Group (n = 40):

Following obtaining their agreement to participate, the Providers will be given a date, time, and venue for his/her participation in the focus group and will meet for one hour. An agenda and script for the conduct of the focus group session will be developed by a trained moderator. The focus groups will be conducted by a member of the research team. Data from the focus group sessions will be analyzed and used to evaluate clinicians' interpretation of patient-reported outcomes (PROs) and acceptability of PRO data in routine clinical care. A formal provider training program will be designed and implemented by a subject matter expert. The focus group session will be repeated at 12 months, with the 12 month administration having an increased emphasis on barriers, facilitators, and value of PROs in clinical care.

Patient Interview Group (n = 100):

Following obtaining agreement to be interviewed, a trained professional interviewer will conduct a one-time, one-hour, semi-structured telephone interview of each subject to better understand patient experiences with HF, the treatment process and quality of life determinants. Two semistructured interviews will be conducted with the first 30 patients who have had left ventricular assist device (LVAD) therapy (of the 100 patients who agreed to be interviewed), before and 12 months after device implantation. The goal of these interviews will be to describe patient experiences with LVAD therapy, examine factors influencing quality of life, and determine whether currently available PRO tools are likely to capture the intended experiences in HF as they relate to LVAD therapy.

PROs/Clinical Data Integration Group (n = 3500):

The patients' electronic medical records will be reviewed and protocol-required information will be obtained. PRO capture will be expanded in a large population of patients across the continuum of HF patients. A plan has been developed that will integrate PRO scores into their medical records. Information will be obtained from 2 instruments (Kansas City Cardiomyopathy Questionnaire (KCCQ12) and NIH Patient Reported Outcomes Measurement Information System (PROMIS)) that are routinely administered as part standard of care. PRO and clinical data will be obtained from electronic medical records of patients seen in the heart failure clinic during the study period. Patient information will be stored in a secure research database. The data will be used to build prognostic models of 1-year survival with favorable quality of life in patients with various forms of heart failure.

No follow-up visits will be required for the PROs/Clinical Data Integration Group. All protocol-required information will be obtained from the subjects' electronic medical records over a period of 3.5 years after enrollment into the study.

Biologic Determinants of Patient Health Status in HF (n = 1000):

Subjects in the Integration Group that meet the inclusion criteria for this subject subset will be contacted in person by the Principal Investigator or his/her delegate. Subjects will be asked if they are willing to provide their blood samples.

Blood samples will be obtained approximately every six months for the duration of the study (i.e., about 4 years). Approximately 40 ml (or 2.71 tablespoons) of venous blood will be obtained on each scheduled blood draw.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants in the Provider Focus Group and Patient Interview Group:

1. Male or female > 18 years of age
2. Ability to understand and provide agreement to participation, which must be obtained prior to initiation of any study procedures
3. Willing and able to comply with the protocol requirements and schedule of evaluations

The Provider Focus Group must meet the following additional criteria:

1. Heart failure providers, including cardiologists, cardiothoracic surgeons, physician assistants, nurse practitioners, nurses, and medical assistants.
2. They are members of the University of Utah and/or Intermountain Medical Center Heart Failure Teams.

The Patient Interview Group must meet the following additional criteria:

1. Documentation of heart failure with reduced ejection fraction (<50%) or heart failure with preserved ejection fraction (>50%)
2. The patient is followed in heart failure clinic at Intermountain Medical Center or the University of Utah
3. Ability to complete PROs, including the KCCQ12 and PROMIS
4. Ability to complete a telephone interview

The PROs/Clinical Data Integration Group must meet the following criteria:

1. Male or female > 18 years of age
2. Documentation of heart failure with reduced ejection fraction (<50%) or heart failure with preserved ejection fraction (>50%)
3. The patient is followed in heart failure clinic at Intermountain Medical Center or the University of Utah
4. No other inclusion criteria are required for this group because study-required information will be obtained from electronic medical records and will not require direct patient contact.

A subset of subjects in this third group (PROs/Clinical Data Integration Group) will be invited to provide a blood sample for the purpose of examining the biological determinants of patient health status in HF, provided they meet the following criteria:

* Age > 18
* Documentation of heart failure with reduced ejection fraction (<50%) or heart failure with preserved ejection fraction (>50%)
* The patient is followed in heart failure clinic at Intermountain Medical Center or the University of Utah
* The patient has no contraindications for blood draws

Exclusion Criteria:

Provider Focus Group:

1. The provider is not interested or is unable to participate in the focus group
2. The Principal Investigator determines that the provider is not eligible for this research study

Patient Interview Group:

1. The patient is not willing to be interviewed
2. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study
3. Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial
4. The Principal Investigator determines that the proposed patient is not eligible for this research study

PROs/Clinical Data Integration Group:

1. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study
2. Other conditions that in the opinion of the Principal Investigator may compromise the quality of the clinical trial
3. The Principal Investigator determines that the proposed patient is not eligible for this research study

A subset of subjects in this third group (PROs/Clinical Data Integration Group) will be invited to provide a blood sample for the purpose of examining the biological determinants of patient health status in HF, except the following:

* Patients who are not interested in providing blood samples
* Patients without heart failure
* Patients with contraindications to blood draws

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All heart failure providers at the Intermountain Medical Center are potential participants in the Provider Focus Group.
  Patients with heart failure who are seen in the HF outpatient clinics at Intermountain Medical Center are potential participants in the Patient Interview Group or the PROs/Clinical Data Integration Group.
Sampling Method: Non-Probability Sample
Enrollment: 3640 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time necessary for PRO completion by patients | 4 years
  It is believed that data entry requirement below 10 minutes is conducive to patient participation and will not interfere with clinic flow. This will me monitored throughout the trial.
Completion rate among eligible patients | 4 years
  PRO completion rate will be closely monitored throughout the study. It is anticipated that the completion rate will exceed 80% and will be sustainable over time.

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah G Kfoury, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Heart Institute, Murray, Utah, United States